CLINICAL TRIAL: NCT00523835
Title: Body Composition, Bone Mineral Density, Insulin Sensitivity and Echocardiographic Measurements in Klinefelter Syndrome
Status: Completed | Type: Observational
Sponsor: University of Aarhus (Other)
Other Study IDs: 20010155
Record Dates: First submitted 2007-08-31; First posted 2007-09-03 (Estimated); Last update posted 2007-09-03 (Estimated); Status verified 2007-08

CONDITIONS: Klinefelter Syndrome; Diabetes; Osteoporosis; Metabolic Syndrome; Cardiovascular Disease
MeSH Terms: conditions — Klinefelter Syndrome; Diabetes Mellitus; Osteoporosis; Metabolic Syndrome; Cardiovascular Diseases

STUDY DESIGN:
Observational Model: Natural History | Time Perspective: Other
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- KS: Patients with Klinefelter syndrome verified by chromosome analysis
- Normal: Normal men Age matched to KS patients

SUMMARY:
Klinefelter syndrome (KS) is the most common sex-chromosome disorder with a prevalence of one in 660 men and is a frequent cause of hypogonadism and infertility. It is caused by the presence of extra X-chromosomes, the most common karyotype being 47,XXY. The phenotype is variable, but the most constant finding is small hyalinized testes, hypergonadotrophic hypogonadism, infertility, eunuchoid body proportion, increased height and learning disabilities. Klinefelter syndrome has been associated with increased prevalence of diabetes, osteoporosis and cardiovascular diseases but the pathogenesis is unknown. Accordingly the aim of the study was to investigate measures of body composition, insulin sensitivity, bone mineral density, echocardiography, as well as biochemical markers of endocrine, metabolic and bone function in KS and an age-matched control group.

ELIGIBILITY:
Inclusion Criteria:

* age above 18 years
* verified KS karyotype (KS patients)

Exclusion Criteria:

* untreated hypothyroidism or hyperthyroidism
* present or past malignant diseases
* clinical liver disease
* treatment with drugs knowing to interfere with glucose homeostasis, fat metabolism or bone modulation (e.g. glucocorticoids)

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 140
Dates: Start 2002-04; Study Completion 2004-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jens S. Christiansen, Professor, Study Chair — Medical department M, Endocrinology and Diabetes, and Medical Research Laboratories, Clinical Institute, Aarhus University Hospital, Denmark; Anders B Bojesen, MD, PhD, Principal Investigator — Medical department M, Endocrinology and Diabetes, and Medical Research Laboratories, Clinical Institute, Aarhus University Hospital, Denmark; Claus H Gravholt, MD, DMsc, PhD, Study Director — Medical department M, Endocrinology and Diabetes, and Medical Research Laboratories, Clinical Institute, Aarhus University Hospital, Denmark
Locations (1):
- Medical department M, Endocrinology and Diabetes, and Medical Research Laboratories, Clinical Institute, Aarhus University Hospital, Aarhus, Denmark

REFERENCES:
- [Result] Bojesen A, Kristensen K, Birkebaek NH, Fedder J, Mosekilde L, Bennett P, Laurberg P, Frystyk J, Flyvbjerg A, Christiansen JS, Gravholt CH. The metabolic syndrome is frequent in Klinefelter's syndrome and is associated with abdominal obesity and hypogonadism. Diabetes Care. 2006 Jul;29(7):1591-8. doi: 10.2337/dc06-0145. PMID 16801584
- [Derived] Overvad S, Bay K, Bojesen A, Gravholt CH. Low INSL3 in Klinefelter syndrome is related to osteocalcin, testosterone treatment and body composition, as well as measures of the hypothalamic-pituitary-gonadal axis. Andrology. 2014 May;2(3):421-7. doi: 10.1111/j.2047-2927.2014.00204.x. Epub 2014 Mar 21. PMID 24659579